CLINICAL TRIAL: NCT04495179
Title: A Phase II, Open-label, Study to Assess the Efficacy, Safety, and Tolerability of AZD4635 in Combination With Durvalumab and in Combination With Cabazitaxel and Durvalumab in Patients Who Have Progressive Metastatic Castrate-Resistant Prostate Cancer (AARDVARC)
Brief Title: A Study of AZD4635 With Durvalumab and With Cabazitaxel and Durvalumab in Patients With mCRPC.
Acronym: AARDVARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8731C00002; 2020-000209-10 (EudraCT Number)
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Progressive Metastatic Castrate-Resistant Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — durvalumab; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: AZD4635 + durvalumab (Experimental): AZD4635 plus durvalumab (Arm A) will consist of participants with mCRPC previously treated with one or more approved NHAs (eg, abiraterone acetate, enzalutamide, apalutamide and/or darolutamide), and one or more taxanes, or participants who are taxane ineligible.
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm B: AZD4635 + durvalumab + cabazitaxel (Experimental): AZD4635 plus durvalumab plus cabazitaxel (Arm B) will consist of participants with mCRPC previously treated with docetaxel and one prior NHA (either abiraterone acetate or enzalutamide but not both (prior apalutamide is not allowed in Arm B).
  Interventions: Drug: AZD4635; Drug: Durvalumab; Drug: Cabazitaxel

INTERVENTIONS:
Drug: AZD4635 — Subjects will receive AZD4635 orally daily
Drug: Durvalumab — Subjects will receive intravenous durvalumab every 4 weeks for Arm A and every 3 weeks for Arm B.
Drug: Cabazitaxel — Subjects will receive intravenous cabazitaxel every 3 weeks
  Arms: Arm B: AZD4635 + durvalumab + cabazitaxel

SUMMARY:
This is a Phase II, international, open-label, two-arm, non-randomised study of AZD4635 in participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a Phase II, international, open-label, two-arm, non-randomised study of AZD4635 in participants with mCRPC. Participants in each arm will be stratified by the presence of measurable soft tissue metastasis (per Response Evaluation Criteria in Solid Tumours [RECIST v1.1]) or bone-only metastasis (per Prostate Cancer Working Group 3 [PCWG3 criteria]). There will be no formal comparisons between treatment arms.

AZD4635 plus durvalumab (Arm A) will consist of 80 participants with mCRPC previously treated with one or more approved new hormonal agent(s) (NHAs) and one or more taxanes or participants who are taxane ineligible.

AZD4635 plus durvalumab plus cabazitaxel (Arm B) will consist of 80 participants mCRPC previously treated with docetaxel and one prior NHA.

As of November 2020, the Sponsor stopped enrolment in Arm A following decisions at the program level, not related to any safety issues. Ongoing participants in Arm A may continue treatment as planned.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. Known castrate-resistant disease.
3. Evidence of disease progression ≤6 months.
4. Body weight >30 kg at screening.
5. Willingness to adhere to the study treatment-specific contraception requirements.
6. Adequate bone marrow reserve and organ function.
7. Adequate organ function for Arm A as demonstrated by all of the following laboratory values:

   * Alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or ≤5 × ULN in the presence of liver metastases.
   * Aspartate aminotransferase (AST) ≤2.5 × ULN if no demonstrable liver metastases or ≤5 × ULN in the presence of liver metastases
   * Total bilirubin (TBL) ≤1.5 × ULN
   * TBL ≤2.0 × ULN in the case of known Gilbert syndrome with normal direct bilirubin
8. Participants in Arm A must have received the following prior therapy:

   * Maximum of 3 lines of therapy in the mCRPC setting
   * Prior therapy with one or more NHAs (eg, abiraterone acetate, enzalutamide, apalutamide, darolutamide) in either hormone-sensitive or hormone-refractory settings
   * Prior therapy with one or more lines of taxanes (eg, docetaxel and/or cabazitaxel)
   * Alternatively, must be taxane-ineligible
   * Prior therapy can be in either the hormone-sensitive or the hormone-refractory setting
9. Adequate organ function for Arm B as demonstrated by all of the following laboratory values:

   * AST and/or ALT ≤1.5 × ULN
   * TBL ≤ ULN
   * TBL ≤2.0 × ULN in the case of known Gilbert syndrome with normal direct bilirubin
10. Participants in Arm B must have received the following prior therapy:

    * Prior docetaxel (taxane) in either hormone-sensitive or hormone-refractory settings
    * Received no prior cytotoxic chemotherapy other than docetaxel for prostate cancer except for estramustine and except adjuvant/neo-adjuvant treatment completed >3 years ago.
    * Prior therapy with only one NHAs (eg, abiraterone acetate or enzalutamide; prior apalutamide is not permitted) for treatment of mCRPC in either hormone-sensitive or hormone-refractory settings.
    * Be suitable to receive concomitant Granulocyte-colony stimulating factor during all cycles of cabazitaxel.
    * Participants who meet inclusion criteria for Arm B will be allocated preferentially to that arm until recruitment to that arm is completed.

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases.
2. There must be no requirement for immunosuppressive doses of systemic corticosteroids for at least 2 weeks prior to study enrollment.
3. History of pneumonitis requiring corticosteroids, second malignancy that is progressing and/or received active treatment ≤3 years before the first dose of study intervention, and hypersensitivity to polysorbate-80 if allocated to cabazitaxel.
4. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases.
5. Creatinine clearance <40 mL/min (calculated by Cockcroft-Gault equation).
6. Prior exposure to immune-mediated therapy including.
7. Ongoing treatment with warfarin (Coumadin).
8. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study intervention.

Ages: 18 Years to 150 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Sweeney, MBBS, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (5):
  - Research Site, Sacramento, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, St Louis, Missouri
  - Research Site, Winston-Salem, North Carolina
- Belgium (2):
  - Research Site, Brasschaat
  - Research Site, Ghent
- France (2):
  - Research Site, Bordeaux
  - Research Site, Villejuif
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00002&attachmentIdentifier=094a199c-bf37-4374-90e2-5f80530bdae1&fileName=D8731C00002_Protocol.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00002&attachmentIdentifier=d3ddec19-8569-41e1-9a0d-d7950c823cc6&fileName=D8731C00002_SAP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00002&attachmentIdentifier=8497cc3d-bcf9-447f-9d24-a712c91a5027&fileName=D8731C00002_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 04-August-2020 to 08-August-2022.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Arm A: AZD4635 + Durvalumab: Participants received AZD4635 Dose A orally daily, and durvalumab Dose B intravenously every 4 weeks.
- Arm B: AZD4635 + Durvalumab + Cabazitaxel: Participants received AZD4635 Dose A orally daily, durvalumab Dose B intravenously (IV) every 3 weeks (Q3W), and cabazitaxel Dose C IV Q3W
Period: Overall Study
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Started | 2 | 28
Completed | 0 | 0
Not Completed | 2 | 28
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Study terminated by sponsor | 0 | 18
Not completed — Death | 0 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all patients who received at least one dose of study treatment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel | Total
Number analyzed (Participants) | 2 | 28 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
  years
    number analyzed (Participants) | 0 | 28 | 28
    (all) |  | 68.0 (8.18) | 68.0 (8.18)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
  Participants
    Male: number analyzed (Participants) | 0 | 28 | 28
    Male | 0 | 28 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk. Population: The number analyzed in the row differs from the overall value as efficacy for low number of participants were not presented.
  Participants
    number analyzed (Participants) | 0 | 28 | 28
    Hispanic or Latino | 0 | 4 | 4
    Not Hispanic or Latino | 0 | 21 | 21
    Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
  Participants
    number analyzed (Participants) | 0 | 25 | 25
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 5 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 19 | 19
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS) in Each Arm Separately to Determine the Efficacy of AZD4635 Plus Durvalumab and of AZD4635 Plus Durvalumab Plus Cabazitaxel in Patients With Metastatic Castrate-resistant Prostate Cancer (mCRPC)
Description: rPFS was defined as the time from first dose to radiographic progression, assessed by the Investigator per RECIST 1.1 (soft tissue) and PCWG3 (Prostate Cancer Working Group 3) criteria [bone] or death from any cause, whichever occurred first.
Time Frame: From first dose to first documented progression or death from any cause (whichever comes first) (approximately 1 year)
Population: Evaluable for efficacy set consisted of dosed patients with a baseline tumour assessment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
months |  | 5.8 [4.2 to NA] — An upper limit for the 95%CI was not calculated because there were not enough events at later times to get a reliable upper CI.

2. Secondary Outcome: rPFS by Adenosine (ADO) Signalling Gene Expression in High and Low Subgroups to Determine the Efficacy of AZD4635 Plus Durvalumab Plus Cabazitaxel in Participants With mCRPC
Description: rPFS was defined as the time from first dose to radiographic progression, assessed by the Investigator per RECIST 1.1 (soft tissue) and PCWG3 criteria (bone) or death from any cause, whichever occurred first.
Time Frame: From first dose to first documented progression or death from any cause (whichever comes first), up to two years
Population: Evaluable for efficacy set consisted of dosed patients with a baseline tumour assessment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk. The analysis of rPFS by ADO was not done.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 27
Participants
  High ADO |  | 14
  Low ADO |  | 13

3. Secondary Outcome: Overall Survival (OS) in Each Arm Separately to Determine the Efficacy of AZD4635 Plus Durvalumab and of AZD4635 Plus Durvalumab Plus Cabazitaxel in Participants With mCRPC
Description: OS was defined as the time from first dose until death due to any cause regardless of whether the participant withdrew from study treatment or received another anti-cancer therapy.
Time Frame: Arm A and B: Every 90 days from the last dose of study drug up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
months |  | NA [7.9 to NA] — This value was not calculated since less than 50% patients died during the study.

4. Secondary Outcome: Number of Participants With Objective Response in Subjects With MCRPC Who Received AZD4635 Plus Durvalumab Plus Cabazitaxel
Description: Confirmed ORR was defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) using overall radiographic response assessed by RECIST v1.1 and PCWG-3 criteria (bone), and was based on a subset of all treated participants with measurable disease at baseline per the site Investigator.
Time Frame: From first dose to first documented progression or death from any cause (whichever comes first), up to two years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Participants |  | 2 [0.88 to 23.50]

5. Secondary Outcome: Number of Participants With Prostate-specifin Antigen (PSA50) Response in Subjects With MCRPC Who Received AZD4635 Plus Durvalumab Plus Cabazitaxel
Description: Confirmed PSA50 response is defined as the proportion of participants who achieved a ≥50% decrease in PSA from baseline to the lowest post-baseline PSA, confirmed by a consecutive PSA at least 3 weeks later and was based on PSA evaluable participants (dosed participants with an abnormal baseline PSA [≥1 ng/mL]).
Time Frame: Arm A: Screening, Day 1 of each cycle up to 11 months (Each cycle was 28 days in length); Arm B: Screening, Day 1 of each cycle up to 11 months (Cycle 1 to Cycle 10 = 21 days, Cycle 11 onwards = 28 days)
Population: PSA evaluable analysis set consisted of dosed participants with an abnormal baseline PSA (=1ng/mL). The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Participants |  | 5 [0.06 to 0.37]

6. Secondary Outcome: Change From Baseline in Worst Pain in the Daily Activities Scales of the Brief Pain Inventory - Short Form (BPI-SF)
Description: "Worst pain" and "Average pain" are 'single question' scores from the BPI short form and may take any value from 0 to 10 (worst outcome). "Interference Pain" is the total score of 7 sub-scores, where each value may take any value from 0 to 10 (worst outcome). The range of the "Interference Score" can be from 0 to 70.
Time Frame: Arm A: Screening, Day 1 of each cycle up to 9 months (Each cycle was 28 days in length); Arm B: Screening, Day 1 of each cycle up to 9 months (Each cycle was 21 days in length)
Population: Full analysis set consisted of all participants who received at least one (non-zero) dose of study treatment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk. Only safety data have been provided.
  None of the 14 participants at Baseline answered the questionnaire at Cycle 1 Day 1. Therefore, related statistics were not derived for this timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Score on a Scale
  Baseline: number analyzed (Participants) | 0 | 14
  Baseline |  | 3.4 (2.44)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 11
  Cycle 2 Day 1 |  | -1.6 (2.94)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 13
  Cycle 3 Day 1 |  | -0.3 (4.40)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 9
  Cycle 4 Day 1 |  | -1.6 (2.88)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 5 Day 1 |  | -2.1 (3.58)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 6 Day 1 |  | -1.9 (3.00)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 7 Day 1 |  | 1.0 (1.85)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 8 Day 1 |  | -1.7 (2.66)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 9 Day 1 |  | -0.2 (2.17)

7. Secondary Outcome: Change From Baseline in Average Pain in the Daily Activities Scales of the Brief Pain Inventory - Short Form (BPI-SF)
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Full analysis set consisted of all participants who received at least one (non-zero) dose of study treatment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk. Only safety data have been provided.
  None of the 14 participants at Baseline answered the questionnaire at Cycle 1 Day 1 and, therefore, related statistics were not derived for this timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Score on a Scale
  Baseline: number analyzed (Participants) | 0 | 14
  Baseline |  | 2.3 (2.09)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 11
  Cycle 2 Day 1 |  | -1.3 (1.19)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 13
  Cycle 3 Day 1 |  | 0.6 (3.15)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 9
  Cycle 4 Day 1 |  | -0.9 (1.27)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 5 Day 1 |  | -1.6 (2.15)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 6 Day 1 |  | -1.4 (1.51)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 7 Day 1 |  | 0.0 (1.41)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 8 Day 1 |  | -0.8 (1.47)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 9 Day 1 |  | -1.2 (0.84)

8. Secondary Outcome: Change From Baseline in Pain Interference in the Daily Activities Scales of the Brief Pain Inventory - Short Form (BPI-SF)
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Score on a Scale
  Baseline: number analyzed (Participants) | 0 | 14
  Baseline |  | 8.0 (8.47)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 11
  Cycle 2 Day 1 |  | 2.5 (13.90)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 13
  Cycle 3 Day 1 |  | 12.3 (18.96)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 9
  Cycle 4 Day 1 |  | 4.9 (12.73)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 5 Day 1 |  | 1.3 (5.19)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 6 Day 1 |  | 2.0 (8.40)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 8
  Cycle 7 Day 1 |  | 8.1 (9.93)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 8 Day 1 |  | 7.2 (13.98)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 9 Day 1 |  | 5.4 (15.16)

9. Secondary Outcome: Number of Participants Who Progressed Based on BPI-SF Item 3
Description: Pain progression was assessed using BPI-SF.
Time Frame: Arm A: Screening, Day 1 of each cycle up to 12 months (Each cycle was 28 days in length); Arm B: Screening, Day 1 of each cycle up to 12 months (Cycle 1 to Cycle 10 = 21 days, Cycle 11 onwards = 28 days)
Population: Full analysis set consisted of all participants who received at least one (non-zero) dose of study treatment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Number; unit: Participants
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Participants |  | 1

10. Secondary Outcome: Change From Baseline in the FACT Advanced Prostate Symptom Indext-6 (FAPSI-6), as Derived From 6 Items, the FAPSI-8 From 8 Items Within the FACT-P and the Prostate Cancer Symptoms (PCS), From the 12 Items in the Prostrate-specific Module of the FACT-P
Description: The Functional Assessment of Cancer Therapy-Prostate (FACT-P) will be used to measure health related quality of life (HRQL) in men with prostate cancer. It consists of 4 subscales (physical, emotional, functional and social/family well-being) plus a 12-item prostate-specific module, the PCS subscale, which highlights concerns specific to participants with prostate cancer. FAPSI-6 is defined as a symptom score made up of 6 items from within the FACT-P (pain [n = 3], fatigue [n = 1], weight loss [n = 1], and concerns about the condition getting worse [n = 1]). Each question in the FACT-P questionnaires has a choice of 5 responses, "Not at all", "A little bit", "Somewhat", "Quite a bit" and "Very much". The scores range from 0 ("Not at all") to 4 ("Very much") for positively phrased questions. Negatively phrased questions have a reverse scoring, from 0 ("Very much") to 4 ("Not at all"). This results in a consistent approach, where higher scores indicate a better quality of life.
Time Frame: as for outcome 6
Population: Full analysis set consisted of all participants who received at least one (non-zero) dose of study treatment. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
  None of the 10 participants at Baseline answered the questionnaire at Cycle 1 Day 1. Therefore, related statistics were not derived for this timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Score on a Scale
  Baseline: number analyzed (Participants) | 0 | 10
  Baseline |  | 16.6 (2.88)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 2 Day 1 |  | 1.9 (1.68)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 9
  Cycle 3 Day 1 |  | -0.7 (5.52)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 4 Day 1 |  | -0.1 (3.34)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 5 Day 1 |  | 0.6 (3.36)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 6 Day 1 |  | 1.5 (1.38)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 7 Day 1 |  | 0.0 (3.92)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 8 Day 1 |  | -1.8 (4.15)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 9 Day 1 |  | -3.0 (4.55)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Investigate the PK of AZD4635 when given in combination with durvalumab, and when given in combination with durvalumab plus cabazitaxel.
Time Frame: Arm A:Cycle 1 to 3, and Cycle 4 onwards, and 90-day follow-up (FU) visit up to 14 months [Each cycle was 28 days in length];Arm B: Cycle 1 to 7 and Cycle 11 onwards, and 90-day FU up to 14 months (Cycle 1 to Cycle 10 = 21 days, Cycle 11 onwards = 28 days)
Population: The pharmacokinetics (PK) analysis set consisted of dosed participants for whom an adequate PK profile was obtained. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Mean (Standard Deviation); unit: nanogram/millilitre (ng/mL)
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 15
nanogram/millilitre (ng/mL) |  | 483.0 (231.1)

12. Secondary Outcome: Terminal Half-life (t1/2λz)
Description: Investigated the PK of AZD4635 when given in combination with durvalumab, and when given in combination with durvalumab plus cabazitaxel.
Time Frame: as for outcome 11
Population: The PK analysis set consisted of dosed participants for whom an adequate PK profile was obtained. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 13
hour (h) |  | 8.87 (4.82)

13. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Zero to the Time of the Last Measurable Concentration (AUClast)
Description: as for outcome 12
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)*nanogram/millilitre (ng/mL)
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 15
hour (h)*nanogram/millilitre (ng/mL) |  | 2787 (1056)

14. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Zero to 24 Hours [AUC(0-24)]
Description: as for outcome 12
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)*nanogram/millilitre (ng/mL)
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 14
hour (h)*nanogram/millilitre (ng/mL) |  | 2874 (1084)

15. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Zero Extrapolated to Infinity (AUCinf)
Description: as for outcome 12
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)*nanogram/millilitre (ng/mL)
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 13
hour (h)*nanogram/millilitre (ng/mL) |  | 3311 (1272)

16. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: as for outcome 12
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 13
Litre |  | 334.6 (254.4)

17. Secondary Outcome: Number of Subjects With Serious and Non-serious Adverse Events
Description: Safety and tolerability of each treatment regimen were assessed in participants with mCRPC.
Time Frame: Arm A: From Screening up to 14 months (Each cycle was 28 days in length); Arm B: From Screening up to 14 months (Cycle 1 to Cycle 10 was 21 days in length, and Cycle 11 onwards was 28 days in length)
Population: The safety analysis set consisted of all participants who received at least 1 dose of study drug. The data for Arm A was not calculated because of only two participants in this arm due to which there will be a patient identification risk.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
Number analyzed (Participants) | 0 | 28
Participants
  Any Adverse Event (AE) |  | 28
  Any AE possibly related to treatment |  | 28
  Any AE possibly related to AZD4635 |  | 23
  Any AE possibly related to Durvalumab |  | 20
  Any AE possibly related to Cabazitaxel |  | 28
  Any AE of CTCAE grade 3 or higher |  | 24
  Any AE of CTCAE grade 3 or higher, possibly related to treatment |  | 20
  Any AE of CTCAE grade 3 or higher possibly related to AZD4635 |  | 9
  Any AE of CTCAE grade 3 or higher possibly related to Durvalumab |  | 9
  Any AE of CTCAE grade 3 or higher possibly related to Cabazitaxel |  | 19
  Any Adverse Event of Special Interest (AESI) for Durvalumab |  | 17
  Any possibly related AESI for Durvalumab |  | 10
  Any AE with outcome = death |  | 2
  Any AE with outcome = death possibly related to treatment |  | 1
  Any Serious Adverse Event (SAE) (including events with outcome = death) |  | 19
  Any SAE (including events with outcome = death) possibly related to treatment |  | 12
  Any SAE leading to discontinuation of AZD4635 |  | 4
  Any SAE leading to discontinuation of AZD4635 possibly related to AZD4635 |  | 1
  Any AE leading to discontinuation of AZD4635 |  | 5
  Any AE leading to dose reduction of AZD4635 |  | 4
  Any AE leading to dose interruption of AZD4635 |  | 15
  Any AE leading to discontinuation of Durvalumab |  | 4
  Any AE leading to dose interruption of Durvalumab |  | 5
  Any AE leading to discontinuation of Cabazitaxel |  | 7
  Any AE leading to dose reduction of Cabazitaxel |  | 4
  Any AE leading to dose interruption of Cabazitaxel |  | 8
  Any other significant AEs |  | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 2 years; Serious and/or other adverse events: From Screening up to 14 months (Each cycle was 28 days in length) for Arm A and from Screening up to 14 months (Cycle 1 to Cycle 10 was 21 days in length, and Cycle 11 onwards was 28 days in length) for Arm B.
Arm/Group | Arm A: AZD4635 + Durvalumab | Arm B: AZD4635 + Durvalumab + Cabazitaxel
All-Cause Mortality (participants affected / at risk) | 2/2 | 7/28
Serious Adverse Events (participants affected / at risk) | 2/2 | 19/28
Other Adverse Events (participants affected / at risk) | 2/2 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: AZD4635 + Durvalumab (N=2) | Arm B: AZD4635 + Durvalumab + Cabazitaxel (N=28)
Abscess neck (Infections and infestations) | 0 (0) | 1
Diverticulitis (Infections and infestations) | 0 (0) | 1
Ureteritis (Infections and infestations) | 0 (0) | 1
Urinary tract infection (Infections and infestations) | 0 (0) | 1
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1
Hypotension (Vascular disorders) | 0 (0) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1
Colitis (Gastrointestinal disorders) | 0 (0) | 1
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1
Nausea (Gastrointestinal disorders) | 0 (0) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1
Vomiting (Gastrointestinal disorders) | 0 (0) | 3
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1
Malaise (General disorders) | 0 (0) | 1
Pyrexia (General disorders) | 0 (0) | 1
Neutrophil Count Decreased (Investigations) | 0 (0) | 1
Acute Post Hemorrhagic Anemia (Blood and lymphatic system disorders) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: AZD4635 + Durvalumab (N=2) | Arm B: AZD4635 + Durvalumab + Cabazitaxel (N=28)
Urinary tract infection (Infections and infestations) | 1 (2) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 1 (4) | 14 (19)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (2) | 5 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 6 (7)
Headache (Nervous system disorders) | 0 (0) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 3 (5)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 14 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 17 (20)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Haematuria (Renal and urinary disorders) | 0 (0) | 5 (7)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 10 (15)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (7)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Amylase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (8)
Weight decreased (Investigations) | 2 (2) | 4 (7)
White blood cell count decreased (Investigations) | 0 (0) | 4 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04495179/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT04495179/SAP_001.pdf